CLINICAL TRIAL: NCT01073150
Title: Tea Tree Oil in the Treatment of Chronic Blepharitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Nahin Geha, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nahin Geha
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Blepharitis
Keywords: Tea Tree Oil; Chronic Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — Tea Tree Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tea Tree Oil — Tea Tree Oil shampoo 0.25% and ointment 5% daily and Tea Tree Oil oily solution 50% once a week for six weeks

SUMMARY:
The purpose of this study is to determine:

* The prevalence of Demodex sp. in chronic blepharitis.
* The efficacy of the treatment of topical Tree Tea Oil in chronic blepharitis for Demodex sp.

DETAILED DESCRIPTION:
Patients with clinical diagnosis of chronic blepharitis were included in this study. A check list of symptoms and an ophthalmologic examination including best corrected visual acuity and biomicroscopy were performed.

Under a slit lamp visualization, three lashes with cylindrical dandruff of each eyelid were epilated by fine forceps. The lashes were immersed in fluorescein dye and examined under a light microscope at a 20-times magnification. The mites were detected based on its morphological characteristics and movement.

The patients with chronic blepharitis who had Demodex were randomly divided in two groups. The treatment group was prescribed lid hygiene with Tea Tree Oil shampoo 0.25% and ointment 5% daily and Tea Tree Oil oily solution 50% once a week - produced by Ophthalmos, São Paulo. The control group used the same posology of placebo similar products.

After six weeks, all subjects underwent the initial clinical and laboratory examination. The symptoms and the quantity of mites (mites/eye) were compared before and after the treatment in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Blepharitis with out treatment previously

Exclusion Criteria:

* Patients under 18 y.o.
* Pregnant woman
* Others Ocular Surface Disease (Severe Dry Eye, Lagoftalmo, Entropium, Ectropium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nahin Geha, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil